CLINICAL TRIAL: NCT01671605
Title: Mechanisms of CKD-Induced Foam Cell Formation
Brief Title: Mechanisms of Chronic Kidney Disease (CKD)-Induced Foam Cell Formation
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Valentina Kon, Principal Investigator, Vanderbilt University
Other Study IDs: 090846
Record Dates: First submitted 2012-08-20; First posted 2012-08-23 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-03

CONDITIONS: Chronic Kidney Disease; Cardiovascular Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CKD not on dialysis: Patients with CKD not on dialysis (CKD III-IV)
- Controls: Controls with normal kidney function (Control)

SUMMARY:
There is currently little understanding of macrophage cholesterol homeostasis and foam cell formation across the spectrum of CKD. We hypothesize that an inverse relationship exist between the severity of CKD and processes underlying foam cell formation, and that the relationship becomes independent of serum lipoprotein levels as renal function declines. We propose to systematically examine scavenger receptors and cholesterol uptake as well as cholesterol transporters and efflux mechanisms in individuals with normal renal function, patients with moderate CKD. We further propose to determine if processed contributing to foam cell formation are related to the plasma lipid profile and if the relationship is modified by co-morbidities, such as diabetes, obesity, systemic inflammation which are common in this population and directly influence vascular integrity. These data will be critically important to understand when the abnormality starts and will provide crucial information.

ELIGIBILITY:
Inclusion Criteria:

Patients with moderate degree of CKD, or patients with advanced CKD or control subjects with intact kidney function

Male or female

All ethnic groups

≥ 18 years and have signed informed consent

Exclusion Criteria:

Pregnancy and current smoking

BMI > 45

Rheumatoid arthritis and systemic lupus erythematosus

History of active or chronic hepatitis B, history of active or chronic hepatitis C, human immunodeficiency virus (HIV)

For moderate CKD subjects: nephrotic syndrome

For control subjects: nephrotic syndrome, patients with estimated GFR < 60 mL/min/1.73 m^2, or proteinuria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CKD not on dialysis (CKD III-IV)
  Controls with normal kidney function (Control)
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2013-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Kon, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Outpatient Dialysis Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CKD Not on Dialysis | Controls
Started | 72 | 31
Completed | 72 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: With or without Chronic Kidney Disease
Groups:
- Total: Total of all reporting groups
Arm/Group | CKD Not on Dialysis | Controls | Total
Number analyzed (Participants) | 72 | 31 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (13.5) | 49.9 (10.6) | 55.9 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 20 | 52
  Male | 40 | 11 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 1 | 16
  White | 56 | 29 | 85
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 72 | 31 | 103
HDL Function [Median (Inter-Quartile Range); unit: Percentage] | 20.8 [16.1 to 23.7] | 26.5 [19.6 to 28.5] | 23.65 [16.1 to 28.5]

OUTCOME MEASURES:

1. Primary Outcome: In Vitro Lipoprotein Functions
Description: Cholesterol efflux. Baseline and outcome measurements are the same. The cholesterol efflux was measured once using HDL isolated from CKD and control patients. There was no intervention,this assessment was performed once in each group. The measurement of cholesterol efflux is performed by an in vitro assay in cultured cells. Cells are loaded with cholesterol and maintained for 72 hours. The media of the cultured cells is then changed and the new media contains HDL from CKD or control patients. In additional cells, no HDL is added. The cells are maintained for 24 hours, and intracellular cholesterol is assessed. The cholesterol efflux represents the amount of cholesterol that was leached by HDL from each of our study groups. Thus, cells not exposed to any HDL will contain the highest intracellular cholesterol content. The amount of cholesterol in cells exposed to CKD HDL or control HDL reflects the efflux capacity of that HDL. This is expressed as percent of cholesterol removed by HDL.
Time Frame: Once, at enrollment
Measure: Median (Inter-Quartile Range); unit: Percentage of cholesterol content
Arm/Group | CKD Not on Dialysis | Controls
Number analyzed (Participants) | 72 | 31
Percentage of cholesterol content | 20.8 [16.1 to 23.7] | 26.5 [19.6 to 28.5]

ADVERSE EVENTS:
Arm/Group | CKD Not on Dialysis | Controls
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/31
Other Adverse Events (participants affected / at risk) | 0/72 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No